CLINICAL TRIAL: NCT00403546
Title: High-Dose Oral Ziprasidone Versus Conventional Dosing in Schizophrenia Patients With Residual Symptoms
Brief Title: High-Dose Oral Ziprasidone Versus Conventional Dosing in Participants With Residual Schizophrenia Symptoms
Acronym: HDZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Donald C. Goff, MD (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-P-001372
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-Dose Ziprasidone (Experimental): Participants with schizophrenia or schizoaffective disorder who remain symptomatic despite treatment with ziprasidone 160 mg/d for at least 3 weeks will be instructed to take ziprasidone oral capsule twice daily added to their regular open-label ziprasidone dose (total of 240 mg/d). After the first week, the study drug will be increased to a total ziprasidone dose of 320 mg/d for 7 weeks.
  Interventions: Drug: Ziprasidone 80-160 mg/d; Drug: Ziprasidone 160 mg/d
- Placebo, Standard Treatment Ziprasidone (Placebo Comparator): Participants with schizophrenia or schizoaffective disorder who remain symptomatic despite treatment with ziprasidone 160 mg/d for at least 3 weeks will be instructed to take matching placebo oral capsule twice daily added to their regular open-label ziprasidone dose of 160 mg/d. After the first week, the matching placebo will be increased to two capsules twice daily and their regular open-label ziprasidone will remain the same (160 mg/d) for 7 weeks.
  Interventions: Drug: Placebo; Drug: Ziprasidone 160 mg/d

INTERVENTIONS:
Drug: Ziprasidone 80-160 mg/d — Participants will be instructed to take one study capsule of ziprasidone orally twice daily (80 mg/d). After the first week, the study drug will be increased to two capsules twice daily (160 mg/d).
  Other Names: Geodon
  Arms: High-Dose Ziprasidone
Drug: Placebo — Participants will be instructed to take one study capsule of matching placebo orally twice daily. After the first week, the matching placebo will be increased to two capsules twice daily.
  Arms: Placebo, Standard Treatment Ziprasidone
Drug: Ziprasidone 160 mg/d — Participants will be taking open-label ziprasidone 80 mg orally twice daily for a total dose of 160 mg/d from at least 3 weeks before randomization to end of study 8 weeks after randomization.
  Other Names: Geodon

SUMMARY:
The primary aims of this study are to assess tolerability of ziprasidone dose escalation to 320 milligrams per day (mg/d) compared to continued standard treatment (placebo) as measured by the Side Effect Checklist, Simpson Angus Scale for Extrapyramidal Symptoms (SAS), Barnes Akathisia Scale (BAS), serum prolactin concentrations, vital signs, electrocardiogram (EKG) and completion rates and to assess whether ziprasidone dose escalation improves overall psychopathology compared to continued standard treatment as measured by the change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score and response rates as defined by a 20% or greater reduction in PANSS total score.

The secondary aims of this study are to assess whether ziprasidone dose escalation improves psychotic symptoms compared to continued standard treatment as measured by the Positive Symptom Subscale of the PANSS, to assess whether ziprasidone dose escalation improves negative symptoms compared to standard treatment as measured by the Negative Symptom Subscale of the PANSS, to assess whether ziprasidone dose escalation improves depressive symptoms compared to continued standard treatment as measured by the Calgary Depression Rating Scale (CDRS), and to assess whether ziprasidone dose escalation improves overall functioning with the Clinical Global Impression - Severity (CGI-S), Clinical Global Impression - Improvement (CGI-I), Global Assessment of Functioning (GAF) and the Schizophrenia Cognition Rating Scale (SCoRS).

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or Schizoaffective disorder, any subtype
* Age 18-65 years
* Treated with ziprasidone at a dose of 160 mg/d for at least 3 weeks with adequate compliance
* Concomitant standing or other medications as needed (except other antipsychotics and those noted as contraindicated in the ziprasidone package insert) are permitted during all treatment phases if they were present at a stable dose for at least 6 weeks prior to the start of initial ziprasidone treatment
* A score of 4 (moderate) or greater on any of the 7 items of the PANSS Positive Symptom Subscale
* Clinical judgment by the investigator that doses higher than 160 mg/day are warranted due to suboptimal clinical outcome despite adequate treatment at that dose
* Participant is judged capable of understanding all relevant risks and potential benefits of the study and has signed informed consent
* Comorbid axis 1 conditions (including anxiety disorders, eating disorders, impulse control disorders) are permitted if they have been stable and have not been a primary focus of treatment over the previous 6 months

Exclusion Criteria:

* Past or current intolerance of ziprasidone side effects
* Presence of significant cardiac disease, including uncompensated congestive heart failure, myocardial infarction within the past 6 months or known history of congenital long QT interval syndrome
* Corrected QT interval (QTc) greater than or equal to 500 milliseconds (msec)
* Serum potassium and magnesium concentrations outside of normal limits.
* Currently taking any medications which may affect cardiac conduction
* Presence of any unstable or untreated medical disorder
* Any history of seizures or seizure disorder other than febrile seizures of childhood
* History of positive hepatitis B surface antigen
* Human immunodeficiency virus (HIV) positive or has diagnosis of acquired immune deficiency syndrome (AIDS)
* Any abnormal laboratory test that is judged to be clinically significant by the investigator
* History of neuroleptic malignant syndrome (NMS), hypersensitivity or allergic response to antipsychotic therapy, including ziprasidone
* History of clozapine treatment for refractory psychotic symptoms
* Alcohol or substance dependence within the past 12 months or abuse within the past 3 months. Any subject with positive urine toxicology or alcohol use that is considered abnormal at baseline.
* Clinically significant suicidal or homicidal behavior or attempts within past 6 months
* Any subject judged by the investigator to present a danger to self or others.
* Women of childbearing potential who are not using adequate contraception (oral contraceptives, barrier methods or who are clearly abstinent)
* Pregnancy or breast-feeding
* Any subject who is judged by the investigator to be unable or unlikely to comply with all study requirements, including adherence with prescribed medication regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, M.D., Principal Investigator — Massachusetts General Hospital
Locations (9):
- United States (9):
  - Medical College of Georgia, Augusta, Georgia
  - Corrigan Mental Health Center, Fall River, Massachusetts
  - Touchstone innovare, Grand Rapids, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - The Lieber Center for Schizophrenia Research - Columbia University, New York, New York
  - Nathan Kline Institute, Orangeburg, New York
  - Duke University - John Umstead Hospital, Butner, North Carolina
  - The Mech Center, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Upon signing informed consent participants not already taking ziprasidone were instructed to start open-label ziprasidone for 3 weeks. Of 131 participants who signed informed consent 75 started ziprasidone and 56 were already on ziprasidone. Those completing open-label and those on ziprasidone were then screened.
Groups:
- Standard Treatment Ziprasidone: Upon signing informed consent participants with schizophrenia or schizoaffective disorder, who were not yet taking ziprasidone could initiate open-label standard treatment ziprasidone (160 milligrams per day [160 mg/d]: 80 mg twice daily) for a minimum of 3 weeks to be eligible for screening to enter the randomized trial. Participants who were already taking standard treatment ziprasidone for 3 weeks or longer at time of enrollment were eligible for screening, as well.
- High-Dose Ziprasidone: Participants with schizophrenia or schizoaffective disorder who remained symptomatic despite treatment with ziprasidone 160 mg/d for at least 3 weeks were instructed to take ziprasidone oral capsule twice daily added to their regular open-label ziprasidone dose (total of 240 mg/d). After the first week, the study drug was increased to a total ziprasidone dose of 320 mg/d for 7 weeks.
- Placebo, Standard Treatment Ziprasidone: Participants with schizophrenia or schizoaffective disorder who remained symptomatic despite treatment with ziprasidone 160 mg/d for at least 3 weeks were instructed to take matching placebo oral capsule twice daily added to their regular open-label ziprasidone dose of 160 mg/d. After the first week, the matching placebo was increased to two capsules twice daily and their regular open-label ziprasidone remained the same (160 mg/d) for 7 weeks.
Period: Signed Informed Consent/Open-Label
Arm/Group | Standard Treatment Ziprasidone | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Started | 131 | 0 | 0
Completed | 103 | 0 | 0
Not Completed | 28 | 0 | 0
Not completed — Withdrew Consent | 6 | 0 | 0
Not completed — Early Termination | 8 | 0 | 0
Not completed — Terminated by Investigator | 9 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Period: Screening Phase
Arm/Group | Standard Treatment Ziprasidone | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Started | 103 | 0 | 0
Completed | 75 (All participants who completed Screening were randomized to the High-Dose and Placebo arms.) | 0 | 0
Not Completed | 28 | 0 | 0
Not completed — Screening Failure | 22 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Terminated Prior to Randomization | 5 | 0 | 0
Period: Randomized Trial
Arm/Group | Standard Treatment Ziprasidone | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Started | 0 (All participants who completed Screening were randomized to the High-Dose and Placebo arms.) | 38 | 37
Completed | 0 | 21 | 21
Not Completed | 0 | 17 | 16
Not completed — Early Terminations | 0 | 17 | 16

BASELINE CHARACTERISTICS:
Population: All participants who entered the Randomized Trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.0) | 41.0 (11.9) | 40.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Events Recorded Based on Ziprasidone Side Effects Checklist During Randomized Trial
Description: Side effects were tracked using the Side Effect Checklist for ziprasidone, which is a well-validated 17 item scale that records the presence or absence of side effects. Total number of side effect events is reported here.
Time Frame: From Baseline up to Week 8
Population: All participants in the randomized trial.
Measure: Number; unit: side effect events
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 37
side effect events | 633 | 588

2. Primary Outcome: Change From Baseline in Simpson Angus Scale for Extrapyramidal Symptoms (SAS)
Description: The SAS is a 10-item testing instrument used to evaluate drug-related extrapyramidal syndromes. The following items are included in the SAS: gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella reflex, tremor, and salivation. Total score ranges from 0 to 40 with a higher score indicating increased severity. A positive change from baseline indicates a worse outcome.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All study participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 37 | 36
units on a scale
  Baseline | 1.5 (2.0) | 1.5 (2.7)
  Change from Baseline at Week 2: number analyzed (Participants) | 32 | 31
  Change from Baseline at Week 2 | 0.44 (1.93) | -0.65 (2.21)
  Change from Baseline at Week 4: number analyzed (Participants) | 26 | 23
  Change from Baseline at Week 4 | 0.46 (2.08) | -0.35 (2.12)
  Change from Baseline at Week 6: number analyzed (Participants) | 22 | 22
  Change from Baseline at Week 6 | 0.59 (3.06) | -0.09 (2.41)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | -0.10 (2.49) | -0.10 (2.02)
Statistical Analysis 1: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Baseline; Test type: Superiority; p = 0.980, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-1.09 to 1.12]
Statistical Analysis 2: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 2; Test type: Superiority; p = 0.033, Mixed Models Analysis; Mean Difference (Net) = 1.02, 95% CI 2-sided [0.08 to 1.95]
Statistical Analysis 3: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 4; Test type: Superiority; p = 0.171, Mixed Models Analysis; Mean Difference (Net) = 0.73, 95% CI 2-sided [-0.32 to 1.77]
Statistical Analysis 4: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 6; Test type: Superiority; p = 0.380, Mixed Models Analysis; Mean Difference (Net) = 0.50, 95% CI 2-sided [-0.62 to 1.62]
Statistical Analysis 5: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 8; Test type: Superiority; p = 0.840, Mixed Models Analysis; Mean Difference (Net) = -0.12, 95% CI 2-sided [-1.32 to 1.08]

3. Primary Outcome: Change From Baseline in the Barnes Akathisia Scale (BAS)
Description: BAS is a rating scale that is administered by physicians to assess the severity of drug-induced akathisia, which is a movement disorder characterized by a feeling of inner restlessness and a compelling need to be in constant motion, as well as by actions such as rocking while standing or sitting, lifting the feet as if marching on the spot, and crossing and uncrossing the legs while sitting. The following subcategories are scored: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness and are rated on a 4-point scale from 0 - 3. In addition, the global clinical assessment of akathisia uses a 6-point scale ranging from 0 - 5. Total score ranges from 0 to 14 with a higher score indicating increased severity. A positive change from baseline indicates a worse outcome.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All participants who had available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 36
units on a scale
  Baseline | 1.2 (2.2) | 1.4 (2.4)
  Change from Baseline at Week 2: number analyzed (Participants) | 33 | 31
  Change from Baseline at Week 2 | 0.00 (2.61) | 0.13 (1.69)
  Change from Baseline at Week 4: number analyzed (Participants) | 26 | 23
  Change from Baseline at Week 4 | -0.27 (2.88) | -0.48 (2.17)
  Change from Baseline at Week 6: number analyzed (Participants) | 22 | 22
  Change from Baseline at Week 6 | -0.95 (2.46) | -0.45 (2.11)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | -0.62 (2.09) | -0.29 (2.15)
Statistical Analysis 1: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Baseline; Test type: Superiority; p = 0.737, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-1.23 to 0.88]
Statistical Analysis 2: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 2; Test type: Superiority; p = 0.764, Mixed Models Analysis; Mean Difference (Net) = -0.14, 95% CI 2-sided [-1.09 to 0.80]
Statistical Analysis 3: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 4; Test type: Superiority; p = 0.642, Mixed Models Analysis; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.82 to 1.32]
Statistical Analysis 4: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 6; Test type: Superiority; p = 0.570, Mixed Models Analysis; Mean Difference (Net) = -0.34, 95% CI 2-sided [-1.50 to 0.83]
Statistical Analysis 5: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 8; Test type: Superiority; p = 0.894, Mixed Models Analysis; Mean Difference (Net) = -0.09, 95% CI 2-sided [-1.34 to 1.17]

4. Primary Outcome: Number of Participants With High and Low Levels in Serum Prolactin Concentration
Description: Blood samples were taken at baseline and Week 8 to measure serum prolactin concentrations. Normal range for females (non-pregnant) is 2-29 nanograms per deciliter (ng/dL) and for males 2-18 ng/dL. Values above the normal range were reported as High and values below the normal range were reported as Low. Reported here is the number of participants with high prolactin concentration and the number of participants with low prolactin concentration.
Time Frame: Baseline, Week 8
Population: All participants with available data at each time point.
Measure: Number; unit: participants
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 37
participants
  High Prolactin at Baseline | 9 | 10
  High Prolactin up to Week 8: number analyzed (Participants) | 21 | 21
  High Prolactin up to Week 8 | 7 | 6
  Low Prolactin at Baseline | 1 | 1
  Low Prolactin up to Week 8: number analyzed (Participants) | 21 | 21
  Low Prolactin up to Week 8 | 1 | 0

5. Primary Outcome: Vital Signs: Systolic and Diastolic Blood Pressure Levels
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured at regular times during the study. Normal SBP is defined as 120 millimeters of mercury (mmHg) or below and normal DBP is defined as 80 mmHg or below. Change from baseline is indicated for each time point. A positive change from baseline indicates and increase in blood pressure and a negative change from baseline indicates a decrease.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 37
mmHg
  SBP Baseline | 123.2 (14.5) | 125.0 (15.3)
  SBP Week 1: number analyzed (Participants) | 38 | 36
  SBP Week 1 | 123.9 (13.58) | 122.3 (15.14)
  SBP Week 2: number analyzed (Participants) | 33 | 31
  SBP Week 2 | 124.5 (14.23) | 124.9 (16.09)
  SBP Week 4: number analyzed (Participants) | 26 | 24
  SBP Week 4 | 124.8 (16.47) | 124.3 (16.92)
  SBP Week 6: number analyzed (Participants) | 22 | 22
  SBP Week 6 | 122.5 (18.63) | 127.3 (13.64)
  SBP Week 8: number analyzed (Participants) | 21 | 21
  SBP Week 8 | 125.1 (16.76) | 121.3 (11.73)
  DBP Baseline | 77.63 (11.49) | 78.43 (9.30)
  DBP Week 1: number analyzed (Participants) | 38 | 36
  DBP Week 1 | 77.18 (9.10) | 76.56 (8.59)
  DBP Week 2: number analyzed (Participants) | 33 | 31
  DBP Week 2 | 79.24 (10.12) | 77.81 (12.16)
  DBP Week 4: number analyzed (Participants) | 26 | 23
  DBP Week 4 | 78.08 (11.36) | 79.17 (10.47)
  DBP Week 6: number analyzed (Participants) | 22 | 22
  DBP Week 6 | 77.73 (14.61) | 82.18 (12.98)
  DBP Week 8: number analyzed (Participants) | 21 | 21
  DBP Week 8 | 79.24 (12.84) | 75.67 (9.70)
Statistical Analysis 1: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; SBP at Baseline; Test type: Superiority; p = 0.599, Mixed Models Analysis; Mean Difference (Net) = -1.82, 95% CI 2-sided [-8.68 to 5.05]
Statistical Analysis 2: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; SBP at Week 1; Test type: Superiority; p = 0.235, Mixed Models Analysis; Mean Difference (Net) = 3.53, 95% CI 2-sided [-2.31 to 9.37]
Statistical Analysis 3: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; SBP at Week 2; Test type: Superiority; p = 0.449, Mixed Models Analysis; Mean Difference (Net) = 2.83, 95% CI 2-sided [-3.80 to 8.57]
Statistical Analysis 4: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; SBP at Week 4; Test type: Superiority; p = 0.301, Mixed Models Analysis; Mean Difference (Net) = 3.64, 95% CI 2-sided [-3.28 to 10.56]
Statistical Analysis 5: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; SBP at Week 6; Test type: Superiority; p = 0.842, Mixed Models Analysis; Mean Difference (Net) = -0.75, 95% CI 2-sided [-8.13 to 6.63]
Statistical Analysis 6: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; SBP at Week 8; Test type: Superiority; p = 0.109, Mixed Models Analysis; Mean Difference (Net) = 6.33, 95% CI 2-sided [-1.43 to 14.09]
Statistical Analysis 7: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; DBP at Baseline; Test type: Superiority; p = 0.741, Mixed Models Analysis; Mean Difference (Net) = -0.80, 95% CI 2-sided [-5.62 to 4.02]
Statistical Analysis 8: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; DBP at Week 1; Test type: Superiority; p = 0.552, Mixed Models Analysis; Mean Difference (Net) = 1.44, 95% CI 2-sided [-3.32 to 6.19]
Statistical Analysis 9: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; DBP at Week 2; Test type: Superiority; p = 0.268, Mixed Models Analysis; Mean Difference (Net) = 2.83, 95% CI 2-sided [-2.18 to 7.84]
Statistical Analysis 10: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; DBP at Week 4; Test type: Superiority; p = 0.719, Mixed Models Analysis; Mean Difference (Net) = 1.02, 95% CI 2-sided [-4.53 to 6.56]
Statistical Analysis 11: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; DBP at Week 6; Test type: Superiority; p = 0.334, Mixed Models Analysis; Mean Difference (Net) = -2.86, 95% CI 2-sided [-8.68 to 2.96]
Statistical Analysis 12: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; DBP at Week 8; Test type: Superiority; p = 0.151, Mixed Models Analysis; Mean Difference (Net) = 4.38, 95% CI 2-sided [-1.61 to 10.37]

6. Primary Outcome: Electrocardiogram (EKG): Number of Participants With an Increase From Baseline to Corrected QT (QTc) Interval >/= 500 Milliseconds (Msec)
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave as determined by electrocardiogram (EKG). The corrected QT Interval (QTc) adjusts the QT interval for heart rate. The number of participants with an increase to QTc interval >/= 500 msec was reported.
Time Frame: 6 hours after dosing of Weeks 1, 2 and 8
Population: All participants with available data at each time point.
Measure: Number; unit: participants
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 34
participants
  Week 1 | 0 | 1
  Week 2: number analyzed (Participants) | 31 | 29
  Week 2 | 0 | 0
  Week 8: number analyzed (Participants) | 21 | 21
  Week 8 | 0 | 0

7. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a medical scale and was used for measuring symptom severity of participants with schizophrenia in this study. Total PANSS score consists of 7 items in the Negative subscale, 7 items in the Positive subscale and 16 items in the General Psychopathology scale. Total PANSS score ranges from 30 to 210. A higher score indicates a worse outcome. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 36
units on a scale
  Baseline | 74.7 (16.1) | 71.9 (12.6)
  Change from Baseline at Week 2: number analyzed (Participants) | 33 | 31
  Change from Baseline at Week 2 | -4.03 (7.65) | -4.16 (9.92)
  Change from Baseline at Week 4: number analyzed (Participants) | 26 | 23
  Change from Baseline at Week 4 | -5.08 (6.91) | -6.87 (9.51)
  Change from Baseline at Week 6: number analyzed (Participants) | 22 | 22
  Change from Baseline at Week 6 | -8.73 (9.48) | -4.32 (11.36)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | -8.62 (7.79) | -5.48 (10.59)
Statistical Analysis 1: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Baseline; Test type: Superiority; p = 0.416, Mixed Models Analysis; Mixed models analysis with random slopes; Mean Difference (Final Values) = 2.77, 95% CI 2-sided [-3.97 to 9.50]
Statistical Analysis 2: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 2; Test type: Superiority; p = 0.854, Mixed Models Analysis; Mean Difference (Net) = 0.37, 95% CI 2-sided [-3.59 to 4.33]
Statistical Analysis 3: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 4; Test type: Superiority; p = 0.406, Mixed Models Analysis; Mean Difference (Net) = 1.95, 95% CI 2-sided [-2.68 to 6.58]
Statistical Analysis 4: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 6; Test type: Superiority; p = 0.256, Mixed Models Analysis; Mean Difference (Net) = -3.01, 95% CI 2-sided [-8.23 to 2.21]
Statistical Analysis 5: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 8; Test type: Superiority; p = 0.642, Mixed Models Analysis; Mean Difference (Net) = -1.37, 95% CI 2-sided [-7.20 to 4.45]

8. Primary Outcome: Percentage of Participants With Response
Description: Response was defined as a reduction in the PANSS total score from baseline by 20% or greater, calculated by first subtracting 30 (the PANSS minimum possible total score). Response rate is the percentage of participants with a response.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All participants with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 33 | 31
percentage of participants
  Week 2 | 24.2 | 38.7
  Week 4: number analyzed (Participants) | 26 | 23
  Week 4 | 23.1 | 60.9
  Week 6: number analyzed (Participants) | 22 | 22
  Week 6 | 36.4 | 31.8
  Week 8: number analyzed (Participants) | 21 | 21
  Week 8 | 33.3 | 42.9

9. Primary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Score
Description: AIMS is a rating scale measuring involuntary movements known as tardive dyskinesia, that sometimes develop as a side effect of long-term treatment with antipsychotic medications. The AIMS score was calculated as the sum of questions 1 through 7 of the AIMS instrument, which includes assessments of involuntary movements in the face, lips, jaw, tongue, upper and lower extremities, and neck/shoulders/hips. Each item is rated on a five-point scale of severity from 0-4 with 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Total scores range from 0 to 28. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 36
units on a scale
  Baseline | 0.6 (1.2) | 1.3 (2.4)
  Change from Baseline at Week 2: number analyzed (Participants) | 33 | 30
  Change from Baseline at Week 2 | 0.00 (1.09) | -0.53 (1.50)
  Change from Baseline at Week 4: number analyzed (Participants) | 26 | 23
  Change from Baseline at Week 4 | 0.46 (1.63) | -0.43 (2.11)
  Change from Baseline at Week 6: number analyzed (Participants) | 22 | 22
  Change from Baseline at Week 6 | 0.55 (1.18) | 0.18 (1.44)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | 0.90 (1.95) | 0.10 (2.07)
Statistical Analysis 1: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Baseline; Test type: Superiority; p = 0.135, Mixed Models Analysis; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.55 to 0.20]
Statistical Analysis 2: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 2; Test type: Superiority; p = 0.262, Mixed Models Analysis; Mean Difference (Net) = 0.44, 95% CI 2-sided [-0.33 to 1.21]
Statistical Analysis 3: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 4; Test type: Superiority; p = 0.209, Mixed Models Analysis; Mean Difference (Net) = 0.58, 95% CI 2-sided [-0.33 to 1.49]
Statistical Analysis 4: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 6; Test type: Superiority; p = 0.950, Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-1.01 to 1.07]
Statistical Analysis 5: Comparison: High-Dose Ziprasidone vs Placebo, Standard Treatment Ziprasidone; At Week 8; Test type: Superiority; p = 0.340, Mixed Models Analysis; Mean Difference (Net) = 0.57, 95% CI 2-sided [-0.61 to 1.76]

10. Primary Outcome: Number of Treatment-emergent Adverse Events During Randomized Trial
Description: Adverse event: any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Serious adverse event (SAE): significant hazard, contraindication, side effect, or precaution, which fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here.
Time Frame: From Baseline up to Week 8
Population: Safety population includes all participants who received at least one dose of study medication.
Measure: Number; unit: adverse events
Groups:
- High Dose Ziprasidone: Participants with schizophrenia or schizoaffective disorder who remained symptomatic despite treatment with ziprasidone 160 mg/d for at least 3 weeks were instructed to take ziprasidone oral capsule twice daily added to their regular open-label ziprasidone dose (total of 240 mg/d). After the first week, the study drug was increased to a total ziprasidone dose of 320 mg/d for 7 weeks.
Arm/Group | High Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 37
adverse events
  Serious Adverse Events | 4 | 3
  Non-serious Adverse Events | 85 | 95

11. Secondary Outcome: Change From Baseline in Positive Subscale Score of PANSS
Description: The PANSS is a medical scale and was used for measuring symptom severity of participants with schizophrenia in this study. Positive symptoms as defined by the American Psychiatric Association refer to an excess or distortion of normal functions and include the following 7 items: delusions, conceptual disorganization, hallucinations, excitement, grandiosity, suspiciousness/persecution and hostility. Score ranges from 7 to 49 with a higher score indicating a worse outcome. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 36
units on a scale
  Baseline | 19.6 (5.5) | 18.2 (5.1)
  Change from Baseline at Week 2: number analyzed (Participants) | 33 | 31
  Change from Baseline at Week 2 | -1.30 (3.25) | -0.90 (3.25)
  Change from Baseline at Week 4: number analyzed (Participants) | 26 | 23
  Change from Baseline at Week 4 | -2.08 (3.19) | -1.57 (3.36)
  Change from Baseline at Week 6: number analyzed (Participants) | 22 | 22
  Change from Baseline at Week 6 | -3.09 (3.75) | -0.91 (3.15)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | -3.24 (3.35) | -1.52 (3.01)

12. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score
Description: The PANSS is a medical scale and was used for measuring symptom severity of participants with schizophrenia in this study. Negative symptoms as defined by the American Psychiatric Association represent a diminution or loss of normal functions and include the following 7 items: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation and stereotyped thinking. Score ranges from 7 to 49 with a higher score indicating a worse outcome. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 36
units on a scale
  Baseline | 18.1 (5.8) | 17.9 (5.3)
  Change from Baseline at Week 2: number analyzed (Participants) | 33 | 31
  Change from Baseline at Week 2 | -0.30 (2.70) | -1.16 (4.66)
  Change from Baseline at Week 4: number analyzed (Participants) | 26 | 23
  Change from Baseline at Week 4 | -1.04 (2.14) | -2.04 (5.80)
  Change from Baseline at Week 6: number analyzed (Participants) | 22 | 22
  Change from Baseline at Week 6 | -1.59 (4.02) | -1.68 (5.45)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | -1.90 (2.98) | -1.52 (5.72)

13. Secondary Outcome: Change From Baseline in the Calgary Depression Rating Scale (CDRS) Total Score
Description: The CDRS was used to assess the level of depression in participants with schizophrenia. The questionnaire consists of 9 questions rated on a 4-point scale from 0 to 3. Total range is 0 to 27 with a higher score indicating a worse outcome. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 37 | 36
units on a scale
  Baseline | 3.8 (3.9) | 4.9 (4.2)
  Change from Baseline at Week 2: number analyzed (Participants) | 32 | 31
  Change from Baseline at Week 2 | -0.72 (3.32) | -1.61 (3.78)
  Change from Baseline at Week 4: number analyzed (Participants) | 26 | 23
  Change from Baseline at Week 4 | 0.19 (3.72) | -1.83 (3.90)
  Change from Baseline at Week 6: number analyzed (Participants) | 22 | 22
  Change from Baseline at Week 6 | -0.32 (3.64) | -2.45 (4.01)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | -0.62 (4.57) | -2.14 (3.84)

14. Secondary Outcome: Change From Baseline in Clinical Global Impression- Severity (CGI-S) Score
Description: CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis. Score ranges from 1 to 7 with a higher score indicating a worse outcome. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 36
units on a scale
  Baseline | 4.1 (0.7) | 4.3 (0.6)
  Change from Baseline at Week 8: number analyzed (Participants) | 20 | 19
  Change from Baseline at Week 8 | -0.25 (0.72) | -0.05 (0.40)

15. Secondary Outcome: Change From Baseline in Clinical Global Impression - Improvement (CGI-I) Score
Description: CGI-I is a 7 point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to baseline. Score ranges from 1 to 7 with a higher score indicating a worse outcome. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 29 | 22
units on a scale
  Baseline | 3.8 (0.5) | 3.9 (0.9)
  Change from Baseline at Week 8: number analyzed (Participants) | 14 | 14
  Change from Baseline at Week 8 | -0.57 (0.94) | -0.43 (0.65)

16. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Score
Description: GAF is a numeric scale used to rate social, occupational, and psychological functioning of participants. Scores range from 100 (extremely high functioning) to 1 (severely impaired). A positive change from baseline indicates an improvement.
Time Frame: Baseline, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 38 | 36
units on a scale
  Baseline | 44.4 (12.3) | 49.0 (14.7)
  Change from Baseline at Week 8: number analyzed (Participants) | 21 | 21
  Change from Baseline at Week 8 | 3.24 (7.76) | 4.86 (11.28)

17. Secondary Outcome: Change in Schizophrenia Cognition Rating Scale (SCoRS) Score
Description: SCoRS is a 20 item interview-based clinical assessment that evaluates cognitive deficits and the degree to which these deficits impair participants' day-to-day functioning. The following cognitive domains are assessed: attention, memory, working memory, language production, reasoning, problem solving, motor skills, and social cognition. Score ranges from 1 to 10 with a higher score indicating a greater degree of impairment. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 8
Population: All participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ziprasidone | Placebo, Standard Treatment Ziprasidone
Number analyzed (Participants) | 37 | 35
units on a scale
  Baseline | 4.9 (1.5) | 4.3 (1.6)
  Change from Baseline at Week 8: number analyzed (Participants) | 20 | 20
  Change from Baseline at Week 8 | -0.75 (0.85) | 0.25 (1.77)

ADVERSE EVENTS:
Time Frame: During open-label phase, screening phase and randomized trial from signing of informed consent up to approximately 12 weeks for participants who initiated ziprasidone as part of the open label phase and 9 weeks for participants who entered directly into the screening phase and randomized trial.
Groups:
- Standard Treatment Ziprasidone Open-label Phase: Upon signing informed consent participants with schizophrenia or schizoaffective disorder, who were not yet taking ziprasidone could initiate open-label standard treatment ziprasidone (160 milligrams per day [160 mg/d]: 80 mg twice daily) for a minimum of 3 weeks to be eligible for screening to enter the randomized trial.
- Standard Treatment Ziprasidone Screening Phase: Participants who had taken standard treatment ziprasidone for 3 weeks or longer were eligible for screening to enter the randomized trial.
- High-Dose Ziprasidone Randomized Trial: Participants with schizophrenia or schizoaffective disorder who remained symptomatic despite treatment with ziprasidone 160 mg/d for at least 3 weeks were instructed to take ziprasidone oral capsule twice daily added to their regular open-label ziprasidone dose (total of 240 mg/d). After the first week, the study drug was increased to a total ziprasidone dose of 320 mg/d for 7 weeks.
- Placebo, Standard Treatment Ziprasidone Randomized Trial: Participants with schizophrenia or schizoaffective disorder who remained symptomatic despite treatment with ziprasidone 160 mg/d for at least 3 weeks were instructed to take matching placebo oral capsule twice daily added to their regular open-label ziprasidone dose of 160 mg/d. After the first week, the matching placebo was increased to two capsules twice daily and their regular open-label ziprasidone remained the same (160 mg/d) for 7 weeks.
Arm/Group | Standard Treatment Ziprasidone Open-label Phase | Standard Treatment Ziprasidone Screening Phase | High-Dose Ziprasidone Randomized Trial | Placebo, Standard Treatment Ziprasidone Randomized Trial
Serious Adverse Events (participants affected / at risk) | 4/131 | 2/103 | 4/38 | 3/37
Other Adverse Events (participants affected / at risk) | 37/131 | 28/103 | 23/38 | 19/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment Ziprasidone Open-label Phase (N=131) | Standard Treatment Ziprasidone Screening Phase (N=103) | High-Dose Ziprasidone Randomized Trial (N=38) | Placebo, Standard Treatment Ziprasidone Randomized Trial (N=37)
Hostility (Psychiatric disorders) | 1 | 1 | 0 | 0
Psychosis (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 1
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychosocial support (Surgical and medical procedures) | 0 | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Asthma (Immune system disorders) | 0 | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment Ziprasidone Open-label Phase (N=131) | Standard Treatment Ziprasidone Screening Phase (N=103) | High-Dose Ziprasidone Randomized Trial (N=38) | Placebo, Standard Treatment Ziprasidone Randomized Trial (N=37)
Hypertension (Vascular disorders) | 12 | 5 | 7 | 5
Constipation (Gastrointestinal disorders) | 4 | 1 | 1 | 4
Tachycardia (Cardiac disorders) | 3 | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 6 | 4 | 2 | 3
Nervousness (Psychiatric disorders) | 3 | 1 | 2 | 3
Paranoia (Psychiatric disorders) | 0 | 1 | 3 | 2
Somnolence (Psychiatric disorders) | 6 | 4 | 6 | 4
Headache (Nervous system disorders) | 3 | 1 | 4 | 2
Malaise (General disorders) | 0 | 0 | 2 | 1
Pain (General disorders) | 0 | 1 | 1 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes